CLINICAL TRIAL: NCT06828705
Title: Establish the First International Database on Semi-quantitative Values Obtained in Scintigraphy With Datscan® in Cadmium-Zinc-Telluride (CZT) Camera (VERITON-CT)
Brief Title: Establish the First International Database on Semi-quantitative Values Obtained in Scintigraphy With Datscan® in Cadmium-Zinc-Telluride Camera
Acronym: DaTBase
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Antoine VERGER, Prinicipal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI206
Record Dates: First submitted 2025-01-31; First posted 2025-02-14 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Neurodegenerative Diseases
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: datscan scintigraphy — Semi-quantitative analysis on Datscan imaging scintigraphy

SUMMARY:
Datscan scintigraphy is a nuclear medicine examination allowing the diagnosis of neurodegenerative pathologies linked to damage to dopaminergic pathways, such as Parkinson's disease (essential for the differential diagnosis of essential tremor).

DETAILED DESCRIPTION:
Datscan scintigraphy is a nuclear medicine examination allowing the diagnosis of neurodegenerative pathologies linked to damage to dopaminergic pathways, such as Parkinson's disease (essential for the differential diagnosis of essential tremor).

There are several types of cameras allowing its performance:

* Conventional Anger cameras and,
* CZT (Cadmium-Zinc-Telluride) semiconductor cameras. At the Nancy University Hospital, the nuclear medicine department has a wide-field Cadmium-Zinc-Telluride camera: VERITON-CT (Spectrum Dynamics). The interpretation of this examination is purely visual.

The objectives are therefore to:

* Create the first international database of semi-quantitative values in 3D scintigraphy with Datscan performed with a VERITON-CT camera.
* Compare this database with another database from a conventional Anger camera (Lyon Nuclear Medicine Department) to show its superiority.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have undergone a Datscan scintigraphy on the VERITON camera in the nuclear medicine department of the Nancy University Hospital and who have an established clinical diagnosis, -Absence of neurodegenerative pathology or Parkinson's disease or Lewy body disease.
* The clinical diagnosis can only be established after two years of clinical follow-up.

Exclusion Criteria:

* Excluded from this research will be the patients opposed to the use of their data, minors, atypical Parkinsonian syndromes,
* patients who died before two years of clinical follow-up,
* patients who had their Datscan examination carried out on a camera other than the VERITON and - patients lost to follow-up.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have undergone a Datscan® scintigraphy on the VERITON-CT camera in the nuclear medicine department of the Nancy University Hospital and who have an established clinical diagnosis, in the absence of neurodegenerative pathology or Parkinson's disease or Lewy body disease
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
To create the first international database of Datscan by camera VERITON-CT. | One day
  Fixation ratio of central gray nuclei of the brain namely, the global striatum, caudate nuclei, putamens

SECONDARY OUTCOMES:
Compare this database with another database from another type of camera (Lyon nuclear medicine team) to show its superiority. | One day
  Identical to the primary evaluation criterion compared to those of the Lyon database.